CLINICAL TRIAL: NCT03705377
Title: Head Start Family and Child Experiences Survey (FACES) 2014-2018
Brief Title: Head Start Family and Child Experiences Survey (FACES 2014)
Acronym: FACES 2014
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Children's Bureau - Administration for Children and Families (Other); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lizabeth Malone, Senior Survey Researcher, Mathematica Policy Research, Inc.
Other Study IDs: 40290A
Record Dates: First submitted 2018-04-03; First posted 2018-10-15 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Head Start Participation
Keywords: child care; child development; child health; child nutrition; child rearing; children; curriculum; early childhood education; families; Head Start; parenting skills; parents; school readiness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head Start children and families: children (2,400), parents (2,400), classrooms/teachers (720), program directors (180), center directors (360), family service staff (168)

SUMMARY:
For nearly two decades, the Head Start Family and Child Experiences Survey (FACES) has been an invaluable source of information on the Head Start program and the children and families it serves. FACES 2014-2018 is the next phase of this important endeavor. Mathematica Policy Research and its partners, Juárez and Associates, Educational Testing Service, and consultants Margaret Burchinal and Martha Zaslow, developed the instruments and data collection procedures to assess the school readiness skills of 2,400 children and survey their parents and Head Start teachers in fall 2014 and spring 2015 (Classroom + Child Outcomes Core) and conduct observations in 720 Head Start classrooms and survey Head Start staff in spring 2015 and spring 2017 (Classroom Core).

DETAILED DESCRIPTION:
The Head Start Family and Child Experiences Survey 2014-2018, or FACES 2014, is the sixth in a series of national studies of Head Start, with earlier studies conducted in 1997, 2000, 2003, 2006, and 2009. It includes nationally representative samples of Head Start programs and centers, classrooms, children and their families. Data from surveys of Head Start program and center directors, classroom teachers, and parents provide descriptive information about program policies and practices, classroom activities, and the background and experiences of Head Start staff and families. Classroom observations are used to assess the quality of Head Start classrooms. Children in the study participate in a direct assessment that provides a rich picture of their school readiness skills at different time points.

FACES 2014 uses a new study design that differs from earlier rounds of FACES in several important ways: (1) it includes larger program and classroom samples, (2) all data are collected in a single program year, (3) the baseline sample of children includes both children enrolled in their first and second year of Head Start, and (4) several special studies are conducted along with the main or Core study to collect more detailed information about a given topic, to study new populations of Head Start programs and participants, and to evaluate measures for possible use in future rounds of FACES. For example, the Family Engagement Plus study in spring 2015 collected information from parents and staff (teachers and family services staff) on family engagement efforts and service provision in Head Start programs. Additional Plus topic modules in spring 2017 gathered information on program functioning from teachers and directors.

The Office of Head Start, the Administration for Children and Families, other federal agencies, local programs, and the public have depended on FACES for valid and reliable national information on (1) the skills and abilities of Head Start children, (2) how Head Start children's skills and abilities compare with preschool children nationally, (3) Head Start children's readiness for and subsequent performance in kindergarten, and (4) the characteristics of the children's home and classroom environments. The FACES study is designed to enable researchers to answer a wide range of research questions that are crucial for aiding program managers and policymakers. Some of the questions that are central to FACES include:

1. What are the demographic characteristics of the population of children and families served by Head Start? How has the population served by Head Start changed?
2. What are the experiences of families and children in the Head Start program? How have they changed?
3. What are the cognitive and social skills of Head Start children at the beginning and end of the program year?
4. Has Head Start program performance improved over time?
5. What are the qualifications of Head Start teachers in terms of education, experience, and credentials?
6. What is the observed quality of Head Start classrooms as early learning environments, including the level and range of teaching and interactions, provisions for learning, emotional and instructional support, and classroom organization? How has quality changed over time? What program- and classroom-level factors are related to observed classroom quality? How is observed quality related to children's outcomes and developmental gains?

ELIGIBILITY:
Inclusion Criteria:

* The Head Start programs participating in FACES 2014 were a probability sample selected from among 2,900 study-eligible programs on the 2012-2013 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be
* In one of the 50 states or the District of Columbia
* Providing services directly to children ages 3 to 5
* Not be in imminent danger of losing its grantee status.

Within those classrooms, eligible classrooms needed to

-have at least one Head Start child enrolled

Exclusion Criteria:

* American Indian and Alaska Native Head Start programs (Region XI) or Migrant and Seasonal Worker Head Start programs (Region XII) were not eligible. Other ACF studies (AI/AN FACES-NCT03842111 and MSHS-NCT03116243) focus on those programs.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head Start children (and their families), Head Start programs, Head Start centers, Head Start classrooms/teachers, Head Start family service staff
Sampling Method: Probability Sample
Enrollment: 5193 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
English proficiency | 1 year
  Children's English language proficiency was assessed during week-long site visits using Preschool Language Assessment Survey (preLAS 2000): Simon Says and Art Show. See Duncan and DeAvila for more information on the scores and technical properties.
  Duncan, S.E., and E. DeAvila. Preschool Language Assessment Survey 2000 Examiner's Manual: English Forms C and D. Monterey, CA: CTB/McGraw-Hill, 1998.
Language-English receptive vocabulary | 1 year
  Indicators of language were assessed during week-long site visits using Peabody Picture Vocabulary Test-Fourth Edition (PPVT-4). See Dunn and Dunn 2006 for more information on the scores and technical properties.
  Dunn, L. M., & Dunn, D. M. Peabody Picture and Vocabulary Test, Fourth Edition. Examiner's Manual and Norms Booklet. Circle Pines, MN: American Guidance Service, 2006.
Language-Expressive vocabulary | 1 year
  Indicators of language were assessed during week-long site visits using Expressive One-Word Picture Vocabulary Test-Fourth Edition (EOWPVT-4 or EOWPVT-4 Spanish-Bilingual Edition). See Martin and Brownell 2011 and Martin 2013 for more information on the scores and technical properties.
  EOWPVT-4: Martin, N., and R. Brownell. "Expressive One-Word Picture Vocabulary Test-4th Edition." Novato, CA: Academic Therapy Publications, 2011.
  EOWPVT-4:SBE: Martin, N. "Expressive One-Word Picture Vocabulary Test-4th Edition: Spanish-Bilingual Edition." Novato, CA: Academic Therapy Publications, 2013.
Language-Spanish receptive vocabulary | 1 year
  Indicators of language were assessed during week-long site visits using Receptive One-Word Picture Vocabulary Test - Fourth Edition (Spanish-Bilingual Edition; ROWPVT-4 SBE). Please see Martin 2012 for more information on the scores and technical properties.
  ROWPVT-4:SBE: Martin, N. "Receptive One-Word Picture Vocabulary Test-Fourth Edition: Spanish-Bilingual Edition." Novato, CA: Academic Therapy Publications, 2012.
Literacy-Letter word knowledge/early writing | 1 year
  Indicators of literacy were assessed during week-long site visits using Woodcock-Johnson III Tests of Achievement-Third Edition/Batería III Woodcock-Muñoz (Spelling, Letter-Word Identification). Please see Woodcock et al. 2001 and Woodcock et al. 2004 for more information on the scores and technical properties.
  English version: Woodcock, R. W., McGrew, K. S. & Mather, N. (2001). Woodcock-Johnson III Tests of Achievement, Itasca, IL: Riverside Publishing, 2001.
  Spanish version: Woodcock, Richard W., Ana F. Munoz-Sandoval, Kevin McGrew, Nancy Mather, and Fred Schrank. Bateria III Woodcock-Munoz. Itasca, IL: Riverside Publishing, 2004.
Literacy-Letter sounds knowledge | 1 year
  Indicators of literacy were assessed during week-long site visits using ECLS-B Letter Sounds. Please see Snow et al. 2007 for more information on the scores and technical properties.
  Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. "Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06)." NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
Mathematics | 1 year
  Indicators of mathematics were assessed during week-long site visits using the Early Childhood Longitudinal Study-Birth Cohort (ECLS-B) preschool mathematics assessment of children's understanding of relative size, ordinal numbers, and pattern matching; number recognition; and the children's ability to count, recognize shapes, add, and solve word problems. Please see Snow et al. 2007 for more information on the scores and technical properties.
  Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. "Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06)." NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
Mathematics | 1 year
  Indicators of mathematics were assessed during week-long site visits using the Woodcock-Johnson III Tests of Achievement-Third Edition/Batería III Woodcock-Muñoz (Applied Problems Test). Please see Woodcock et al. 2001 and Woodcock et al. 2004 for more information on the scores and technical properties.
  English version: Woodcock, R. W., McGrew, K. S. & Mather, N. (2001). Woodcock-Johnson III Tests of Achievement, Itasca, IL: Riverside Publishing, 2001.
  Spanish version: Woodcock, Richard W., Ana F. Munoz-Sandoval, Kevin McGrew, Nancy Mather, and Fred Schrank. Bateria III Woodcock-Munoz. Itasca, IL: Riverside Publishing, 2004.)
Children's physical health | 1 year
  Indicators of physical well-being were assessed by weighing (using kilograms) and measuring children's height (using centimeters), and using these measurements to calculate Body Mass Index (BMI)
General health status | 1 year
  Indicators of physical well-being were assessed by parent report to a survey item on if child's health is excellent, very good, good, fair, or poor
Executive function | 1 year
  Indicators of executive function were assessed by a pencil-tapping task that requires the child do the opposite of what the assessor says (that is, tap one time when the assessor taps two times and tap two times when the assessor taps one time). Pencil Tapping provides an objective assessment of children's self-regulation, particularly inhibitory control and working memory.
  See Blair 2002 for example for more information on the task.
  Blair, C. "School Readiness: Integrating Cognition and Emotion in a Neurobiological Conceptualization of Children's Functioning at School Entry." American Psychologist, vol. 57, 2002, pp. 111-127.
Social-emotional development | 1 year
  Indicators of social-emotional development were assessed using teacher report of several items on children's positive and problem behaviors. Please see the FACES 2014 User's Manual (Kopack Klein et al. 2017) for more information on the scores and technical information.
  Kopack Klein, A., B. Lepidus Carlson, N. Aikens, A. Bloomenthal, J. West, L. Malone, E. Moiduddin, M. Dang, M. Hepburn, S. Skidmore, S. Bernstein, A. Kelly, F. Hurwitz, A. Edwards, H. Zhou, and G. Lim. "Head Start Family and Child Experiences Survey (2014) User's Manual." Report submitted to the U.S. Department of Health and Human Services, Administration for Children and Families, Office of Planning, Research, and Evaluation. Washington, DC: Mathematica Policy Research, 2017.
Social-emotional development-cognitive/social behaviors | 1 year
  Indicators of social-emotional development were assessed using assessor report children's cognitive/social behaviors during the assessment time, using the Leiter-R Examiner Ratings. The Leiter-R comprises eight subscales that examine children's approach to the assessments, their engagement with the materials, and their ability to attend to and regulate their physical and emotional responses during the assessment tasks. Please see Roid and Miller 1997 for more information on the scores and technical properties.
  Roid, G.H., and L.J. Miller. Leiter International Performance Scale Revised, Examiner Rating Scale (Leiter-R). Lutz, FL: Psychological Assessment Resources, Inc., 1997.
Social-emotional development - Approaches to learning | 1 year
  Indicators of social-emotional development were assessed using teacher report of approaches to learning using the Early Childhood Longitudinal Study - Kindergarten Class of 1998 (ECLS-K). The items assess a child's motivation, attention, organization, persistence, and independence in learning. Please see U.S. Department of Education 2002 for more information on the scores and technical properties.
  U.S. Department of Education, National Center for Education Statistics. "Early Childhood Longitudinal Study-Kindergarten Class of 1998-99 (ECLS-K), Psychometric Report for Kindergarten through First Grade." NCES 2002-05. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2002.
Classroom quality-teacher child interactions | One-day observation in March-May 2015, March-May 2017
  Indicators of classroom quality were assessed using the the PreK Classroom Assessment Scoring System. The Pre-K CLASS assesses the qualities of interactions between teachers and students in classrooms and measures aspects of interactions related to children's early academic achievement and social competencies. Please see Pianta et al. 2008 for more information on the scores and technical properties.
  Pianta, Robert, K. LaParo, and B. Hamre. The Classroom Assessment Scoring System Pre-K Manual. Charlottesville, VA: University of Virginia, 2008.
Classroom quality-global classroom environment | One-day observation in March-May 2015, March-May 2017
  Indicators of classroom quality were assessed using a shortened form of the Early Childhood Environment Rating Scale-Revised (ECERS-R), a global rating of classroom quality based on structural features of the classroom (Harms et al. 2005). The items in the short form represent the strongest 21 items identified by researchers in a large-scale study (Clifford et al. 2005). Please see Harms et al. 2005 and Clifford et al. 2005 for more information on the scores and measure technical properties.
  Harms, T., R.M. Clifford, and D. Cryer. Early Childhood Environment Rating Scale: Revised Edition. New York: Teachers College Press, 2005.
  Clifford, Richard, Oscar Barbarin, Florence Chang, Diane M. Early, Donna Bryant, Carollee Howes, Margaret Burchinal, and Robert Pianta. "What Is Pre-Kindergarten? Characteristics of Public Pre-Kindergarten Programs." Applied Developmental Science, vol. 9, no. 3, 2005, pp. 126-143.

CONTACTS AND LOCATIONS:
Overall Officials: Lizabeth Malone, Ph.D., Study Director — Mathematica Policy Research; Nikki Aikens, Ph.D., Principal Investigator — Mathematica Policy Research; Louisa Tarullo, Ed.D., Principal Investigator — Mathematica Policy Research
Locations (1):
- Mathematica Policy Research, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
The FACES Study team will prepare restricted-use data files and documentation so that future researchers may use the data to replicate findings and explore new areas of inquiry.
Supporting Information: Study Protocol
Time Frame: Data are currently available for fall 2014-spring 2015. Data for spring 2017 will become available within 2 years of the end of the study and will remain on ResearchConnections.org.
Access Criteria: Applications for access to restricted-use data file include completing and adhering to a User Agreement.
URL: https://www.researchconnections.org/childcare/studies/36643

REFERENCES:
- See also: To learn more about FACES and access reports/products, please visit the FACES ACF website. — https://www.acf.hhs.gov/opre/research/project/head-start-family-and-child-experiences-survey-faces